CLINICAL TRIAL: NCT00067496
Title: Modafinil in the Treatment of Fatigue in Post-Polio Syndrome
Brief Title: Modafinil to Treat Fatigue in Post-Polio Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030276; 03-N-0276
Record Dates: First submitted 2003-08-20; First posted 2003-08-21 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2005-05

CONDITIONS: Postpoliomyelitis Syndrome
Keywords: Pain; Weakness; Depression; Poliomyelitis; Sleep Apnea; Post-Polio Syndrome; PPS
MeSH Terms: conditions — Postpoliomyelitis Syndrome; Pain; Asthenia; Depression; Poliomyelitis; Sleep Apnea Syndromes | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
This study, conducted at the Walter Reed Army Medical Center, the National Rehabilitation Hospital, and the National Institutes of Health, will examine whether the drug Modafinil can decrease fatigue in patients with post-polio syndrome. Many people who have had polio develop weakness and severe fatigue several years after their recovery from the acute disease. Modafinil is approved by the Food and Drug Administration to improve wakefulness in patients with narcolepsy (disease in which patients have excessive daytime sleepiness) and has been used to treat patients with fatigue related to other medical conditions, such as multiple sclerosis. This study will compare the effects of two doses of Modafinil and of a placebo (a pill with no active ingredient) on fatigue in patients with post-polio syndrome.

Patients who develop fatigue, weakness, muscle pain or atrophy, and functional loss at least 15 years after recovering from polio and whose symptoms cannot be attributed to another cause may be eligible for this study. Candidates will be screened with a medical history, physical and neurological examinations, fatigue rating scales, electrocardiogram, blood and urine tests, drowsiness and depression evaluations, and an electroymogram (EMG) to diagnose nerve or muscle problems. For the EMG, electrodes (small metal discs) are taped to the skin and a needle is inserted into a muscle to record the electrical activity.

Candidates will also undergo a sleep study to exclude abnormal sleep patterns as the cause of the fatigue. For this study, patients stay overnight at the NIH hospital. Electrodes are placed on the throat, on a finger, and on the chest (for an electrocardiogram), and a respiratory belt is placed around the chest-abdomen area. During sleep (from 10:30 p.m. to 6 a.m.), brain waves, eye and leg movements, muscle tone, respiration, and heart rate are recorded. Beginning at 8 a.m. the following morning, the patient takes 20-minute naps to measure the level of daytime sleepiness, using a recording technique similar to that of the all-night study. When five naps are completed, the sleep study ends. Candidates may also undergo a lumbar puncture (spinal tap) to check for certain chemicals in the spinal fluid that might be related to fatigue and to look for possible causes of post-polio syndrome. This procedure is optional. For the lumbar puncture, a local anesthetic is given and a needle is inserted in the space between the bones in the lower back where the cerebrospinal fluid circulates below the spinal cord. A small amount of fluid is collected through the needle.

Patients enrolled in the study will complete a sleep diary during the entire study period. They will be randomly assigned to one of two treatment groups-Modafinil or placebo-for 6 weeks, followed by a 2-week washout period with no medication, and then a crossover phase, in which patients who took Modafinil for the first 6 weeks now take placebo, and those who took placebo now take Modafinil.

At the first study visit, patients will be given a supply of study medication and have blood drawn. They will take one pill twice a day during both study phases. In both study phases, evaluations will be done 3 and 6 weeks after starting the medication. The evaluations include filling out the same forms completed at the screening visit, a review of drug side effects, and a review of medical problems since the last study visit. At the 6-week visit, blood is also drawn.

DETAILED DESCRIPTION:
The main objective of this study is to determine if the drug Modafinil is effective in the treatment of fatigue in patients with post-polio syndrome (PPS). PPS is a motor neuron disease experience by more than 400,000 Americans, characterized by new weakness and intense fatigue. The cause of fatigue, the most common and disabiling symptom in these patients, is unknown and there is no effective treatment. In the present study, selected PPS patients will be randomized to receive two different doses of Modafinil or placebo. After six weeks, the patients will enter a two-week wash out period, and then will be crossed over to the other arm. The sample size has been powered to reflect a significant difference in the scales of fatigue. Secondary exploratory studies will include investigation of sleep patterns as a cause contributing to fatigue and a search for upregulation of fatigue-associated cytokines in the patient's serum and CSF.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will have to meet the clinical criteria for the diagnosis of PPS, have fatigue as a major complaint, and be 18 years or older, of either sex.

EXCLUSION CRITERIA:

Sensitivity to modafinil.

A score of 34 or below on the FSS.

Suffer from depression (BDI-II score of 31 or higher) severe enough to compound the fatigue evaluation.

Another general medical condition that might produce fatigue to a sufficient degree to compound and confuse the assessment of fatigue due to PPS.

Use of a drug known to cause a clinically significant interaction with modafinil.

Presence of sleep disorder suggested by Epworth Sleepiness Scale (score of 18 or higher), patient history, sleep diary or polysomnogram.

Pregnancy .

Breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-08; Study Completion 2006-08

PRIMARY OUTCOMES:
Ascertain whether modafinil is of any benefit in alleviating the fatigue of Post-Polio Syndrome.

SECONDARY OUTCOMES:
Determine if fatigue reduction, correlates with improvement in quality of life of subjects with Post-Polio Syndrome. Investigate the pathophysiology of Post-Polio Syndrome by the study of serum and CSF for evidence of inflammatory markers.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Nollet F, Beelen A, Prins MH, de Visser M, Sargeant AJ, Lankhorst GJ, de Jong BA. Disability and functional assessment in former polio patients with and without postpolio syndrome. Arch Phys Med Rehabil. 1999 Feb;80(2):136-43. doi: 10.1016/s0003-9993(99)90110-7. PMID 10025486